CLINICAL TRIAL: NCT04460963
Title: Role of Adrenomedullin in Leukemic Endosteal/Vascular Niches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AML2220
Record Dates: First submitted 2020-06-25; First posted 2020-07-08 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: adrenomedullin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Adrenomedullin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological evaluation (Other): Adrenomedullin evaluation at diagnosis at first CR and 1 year of follow-up
  Interventions: Other: Adrenomedullin

INTERVENTIONS:
Other: Adrenomedullin — Adrenomedullin sample evaluation

SUMMARY:
The present study will be divided into 5 phases:

1. Collection of bone marrow and peripheral blood (PB) samples from AML patients at diagnosis;
2. Measurement of Midregional Proadrenomedullin (MR-proADM) plasma concentrations with an Immunoluminometric Assay of newly diagnosed AML patients not affected by concomitant cardiovascular disease or sepsis.
3. Analysis of exosomes and microvesicles derived from PB and bone marrow samples of AML patients and culture media collected from AML samples stimulated with ADM and/or ADM (22-52)
4. Study of adrenomedullin system in leukemic stem cells (CD44+/CD38-/CD31+/Lin-) in order to define a correlated expression of ADM and ADM receptors (RAMPs, PAM) with adhesion molecules (CD31, CD38, CD44s, CD44v6), cell cycle regulatory proteins (p21, p27) and genes or molecules involved in the hematopoietic differentiation process (Cul5, CD11b, CD11c, CD66, CD14, CD15, PML-RARα)
5. In vitro evaluation of ADM activity in the growth, maturation and trans-endothelial migration of blasts and/or fusion of leukemic cells with endothelial cells. To do this, leukemic cells will be alternatively cultured by using in vitro models of endosteal and vascular niches.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with new diagnosis of primary or secondary AML.
2. Participant is willing and able to give signed written informed consent according to ICH/EU/GCP and national local laws.
3. Male or Female, aged >18 years.

Exclusion Criteria:

1. Patients affected by concomitant cardiovascular disease , such as essential hypertension (any grade), chronic renal failure (creatinine>1.5 mg/dL), heart failure (any NYHA class), and peripheral arterial occlusive diseases, or sepsis.
2. Patients affected by HIV, B or C hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of therapeutic potential of ADM inhibition on leukaemia stem cells | at 1 year
  Rate estimation of the in vitro arrest of leukemic blasts proliferation by ADM inhibition.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - As Dell'Alto Adige, Ospedale Centrale Di Bolzano - Ematologia E Centro Trapianto Midollo Osseo, Bolzano
  - U.O. Oncoematologia IOV, Castelfranco Veneto
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - Ematologia, San Giovanni Rotondo
  - Uo Ematologia - Azienda Ulss N.2 Marca Trevigiana, Treviso